CLINICAL TRIAL: NCT01061268
Title: A Randomized Clinical Evaluation Pilot Study of the Efficacy of Blink® Tears Lubricant Eye Drops for the Relief of Dry Eye Symptoms Following Implantation of Tecnis® Multifocal Introcular Lens
Brief Title: A Clinical Evaluation Pilot Study of the Efficacy of Blink® Tears Lubricant Eye Drops for the Relief of Dry Eye Symptoms Following Implantation of Tecnis® Multifocal Introcular Lens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMF-001
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: Relief of dry eye symptoms following implantation of TMF IOL
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BLINK™ tears (Experimental)
  Interventions: Drug: Blink® Tears Lubricant Eye Drops
- No topical artificial tear (No Intervention)
  Interventions: Drug: No topical artificial tear

INTERVENTIONS:
Drug: No topical artificial tear — 40 patients randomized to not using a topical artificial tear.
  Arms: No topical artificial tear
Drug: Blink® Tears Lubricant Eye Drops — Blink® Tears Lubricant Eye Drops
  Arms: BLINK™ tears

SUMMARY:
To evaluate the safety and efficacy of BLINK™ tears compared with NO topical artificial tear use in improving subject's visual performance and reduce ocular symptoms of discomfort in subjects who have undergone cataract surgery implanted with a Tecnis™ diffractive multifocal intraocular lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 21 years of age or older
* Written, informed consent and HIPPA Authorization
* Has 20/40 or better best corrected visual acuity in the surgical eye at the Day 1 post-op visit (Visit 3)
* Has undergone cataract surgery in only one eye and has received a Tecnis multi-focal intraocular lens in the study eye.
* Patients not currently using any artificial tears regularly, or using low viscosity tears for symptom relief (Refresh Tears, Visine Tears, Tears Naturelle, etc.)
* Likely to complete the entire course of the study.

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
* Subjects with diabetes mellitus
* Uncontrolled systemic or ocular disease
* History of ocular trauma or prior ocular surgery
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
* Contact lens usage within 6 months for PMMA contacts lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft contact lenses
* A subject whose best-corrected visual acuity is worse than 20/40 in their surgical eye
* A subject with any UNCONTROLLED systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
* A subject that required the use of any artificial tear supplements, vasoconstrictor and/or redness reliever ocular drops 28 days prior to or during the study period
* A subject that required the use of cyclosporine ocular drops 3 months prior to or during the study period
* A subject with active ocular inflammation or corneal edema beyond what is expected on Day 1 after cataract surgery in the study eye
* A subject with a history of conjunctivitis or ocular infection in the study eye within the past 3 months, or a history of kerato-refractive surgery in the study eye within the past 6 months of entry in to the study
* A subject that has punctual plug(s), intracanalicular plug(s) or a history of punctual cautery in the study eye

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of BLINK™ tears | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bloomenstein, M.D., Principal Investigator — Schwartz Laser Eye Center
Locations (1):
- Schwartz Laser Eye Center, Scottsdale, Arizona, United States